CLINICAL TRIAL: NCT06722027
Title: Compassion-Centered Spiritual Health Interventions for Teams (CCSH-TI) With Faculty and Staff
Brief Title: CCSH (Compassion-Centered Spiritual Health) for Teams
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jennifer Mascaro, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00006109; 1R34AT012509-01A1 (NIH)
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Health Behavior
Keywords: Behavioral Intervention; Healthcare provider burnout
MeSH Terms: conditions — Health Behavior | interventions — Therapeutics; Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a longitudinal, randomized pilot study of 80 employees working in inter-professional oncologic teams. Employees will be randomized by team (using a random number generator in Microsoft Excel) to receive CCSH-TI or to a TAU "treatment as usual" (TAU) group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CCSH-TI Group (Experimental): 4-session intervention of 60- minutes each delivered every other week by healthcare chaplains to mixed-role inter-professional teams that includes mindfulness and compassion-based approaches to bolster resilience, compassion for self and others, and psychological safety.
  Interventions: Behavioral: Compassion Centered Spiritual Health Team Intervention (CCSH-TI)
- TAU (treatment as usual) group (Active Comparator): Participants in this group will have access to all well-being resources and activities available to them as employees.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Compassion Centered Spiritual Health Team Intervention (CCSH-TI) — Delivered to healthcare teams by spiritual health clinicians proficient in group facilitation. It is composed of 4 sessions delivered every other week and lasting 60 minutes each.
  CCSH-TI sessions teach participants to attune to their interpersonal relationships; acknowledge and allow difficult emotions; and access compassion. It also provides psychoeducation about skillful coping strategies. Each session consists of didactic material about team norms and safety, a feeling check-in, facilitated group discussions about social connection and professional team building, and meditations to promote mindfulness, to cultivate a feeling of being nurtured, and to access compassion for self and others. CCSH-TI is delivered to healthcare teams by spiritual health clinicians proficient in group facilitation.
  Other Names: CCSH-TI
  Arms: CCSH-TI Group
Behavioral: Treatment as Usual — TAU refers to the current buffet of wellness and professional development activities that are available to employees at the Winship Cancer Institute.
  Other Names: TAU; Standard of Care
  Arms: TAU (treatment as usual) group

SUMMARY:
Emory Spiritual Health has developed a Compassion-Centered Spiritual Health group-based intervention, called CCSH Interventions for Teams, and are enrolling staff and providers into the groups in this randomized study design. The groups will meet once every other week for 60 minutes for 8 weeks (4 sessions total).

The investigators will evaluate the feasibility and acceptability of this novel team-based intervention that includes mindfulness and compassion-based approaches with mixed-role oncology teams. Employees (n = 80; nurses, advanced practice providers (APPs), physicians, staff) working at an NCI- designated Comprehensive Cancer Center will be randomized by team (8-12 employees/group) to Compassion Centered Spiritual Health Team Intervention (CCSH-TI) or TAU (Treatment as Usual) group. The research objective is to evaluate the feasibility and acceptability of CCSH-TI, and to develop and validate a novel, low-burden ambulatory assessment "toolkit" to improve the measurement of psychological safety and burnout.

DETAILED DESCRIPTION:
Current interventions to reduce provider burnout are only minimally effective. To overcome the barriers to achieving success in burnout prevention interventions, the investigators propose Compassion Centered Spiritual Health Team Intervention (CCSH-TI), a 4-session intervention delivered by healthcare chaplains to mixed-role interprofessional teams that includes mindfulness and compassion-based approaches to bolster resilience, compassion for self and others, and psychological safety. The research team will conduct a mixed-method feasibility and acceptability study of CCSH-TI with mixed-role oncology teams. Employees (n = 80; nurses, advanced practice providers (APPs), physicians, staff) working at an NCI-designated Comprehensive Cancer Center will be randomized by team (8-12 employees/group) to CCSH-TI or to TAU (Treatment as Usual) group, who has access to all well-being resources and activities available to them as employees. Self-report surveys and focus group discussions will be used to evaluate the feasibility and acceptability of CCSH-TI. The investigators will also collect self-report surveys, ecological momentary assessments (EMA), and the electronically activated recorder (EAR) data at 3 timepoints (before CCSH-TI (T1), immediately after completion of CCSH-TI (T2), and 12-weeks after completion (LT), and characterize data completion to evaluate the feasibility of data collection methods for a future randomized control trial. Informed consent will be obtained from study participants in-person. The duration of the study will be 22-23 weeks (from consent to completion of data collection).

ELIGIBILITY:
Inclusion Criteria:

* Full-time employees working in oncology teams at Winship Cancer Institute;
* Employees working in intensive care at Emory University St. Joseph hospital.

Exclusion Criteria:

* Less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible employees who enroll and are willing to be randomized | BaselineI (T1), immediately post-intervention (T2), and 12-weeks post-intervention (LT)
  Proportion of eligible employees (all, and according to license, sex/gender, race/ethnicity) who enroll and are willing to be randomized.
Number of participants that attended and completed the three assessment timepoints | BaselineI (T1), immediately post-intervention (T2), and 12-weeks post-intervention (LT)
  Number of participants that attended and completed the three assessment timepoints
Retention rates at three assessment timepoints | BaselineI (T1), immediately post-intervention (T2), and 12-weeks post-intervention (LT)
  Retention rates will be assessed at three assessment timepoints
Satisfaction score | Immediately post-intervention (T2), and 12-weeks post-intervention (LT)
  The investigators will administer a satisfaction questionnaire that includes 5 questions. Total possible score ranges from 5-25. With higher score correlating with better study outcome.
Perceived credibility score | Immediately post-intervention (T2), and 12-weeks post-intervention (LT)
  The investigators will assess perceived credibility with a questionnaire that includes 5 questions. Each question is scores from 1 to 8 with a total possible score range of 5-40. Higher score correlates with better study outcome.
Perceived intervention benefit | Immediately post-intervention (T2), and 12-weeks post-intervention (LT)
  The investigators will assess perceived benefit with a questionnaire that includes 18 questions, to be answered with a 7-point scale. Total possible score ranges from 18 to 126. Higher score correlates with better study outcome.
Acceptability of wearing the Electronically Activated Recorder (EAR) | BaselineI (T1), immediately post-intervention (T2), and 12-weeks post-intervention (LT)
  After the T1, T2, and LT assessments, participants will complete the EAR Experiential Questionnaire, a self-report measure that assesses the acceptability of wearing the EAR. Questions focus on participants' comfort with wearing the EAR, whether the EAR impeded daily activities, whether the EAR changed their behaviors or others' behaviors, and how typical were the days that the EAR was worn. Each question is rated on a Likert scale (1 "not at all" - 5 "a great deal"). Higher score correlates with better outcome.
Number of EMA dropouts | BaselineI (T1), immediately post-intervention (T2), and 12-weeks post-intervention (LT)
  Number of EMA dropouts will be collected
Percentage (%) of items completed using EMA | BaselineI (T1), immediately post-intervention (T2), and 12-weeks post-intervention (LT)
  Percentage of items completed using EMA will be assessed.

SECONDARY OUTCOMES:
Change in Agency for Healthcare Research and Quality's TeamSTEPPS ® Teamwork Perceptions Questionnaire (T-TPQ) score | BaselineI (T1), immediately post-intervention (T2), and 12-weeks post-intervention (LT)
  Measures perceptions of team function with the administration of the Team Structure and Mutual Support subscales (14 items total). Total possible score ranges from 1-14 with higher scores indicating better outcome.
Change in Psychological safety scale score | BaselineI (T1), immediately post-intervention (T2), and 12-weeks post-intervention (LT)
  Includes subscales measuring psychological safety with leaders, peers, and within the team (19 items). Total possible score ranges from 1-19 with higher scores indicating better outcome.
Change in Professional Fulfillment Index Score | BaselineI (T1), immediately post-intervention (T2), and 12-weeks post-intervention (LT)
  Measures Professional fulfillment and burnout, and has demonstrated sensitivity to change in intervention studies (16 items). Total possible score ranges from 1-16 with higher scores indicating better outcome.
EMA (ecological momentary assessment) questionnaire score | BaselineI (T1), immediately post-intervention (T2), and 12-weeks post-intervention (LT)
  The 3-day ambulatory questionnaire asks participants whether the ecological momentary assessment (EMA) impeded daily activities or changed their behaviors, rated on a Likert scale (1 "not at all" - 5 "a great deal"). Higher score correlates with better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Mascaro, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Emory University St. Joseph hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
The research team will share the molar and behavioral codebooks by uploading them to the Open Science Framework (OSF) EAR Repository, a publicly asses-sable collaborative repository of EAR, a resource co-maintained by a member of the research team (Kaplan). The investigator will share summarized rates of accrual, retention, intervention attendance, and self-reported data (mean, standard deviation, and range) at all 3 time-points.
  Access will not be controlled or monitored; it will be made available by the data repository based on approval guidelines maintained by the repository itself.
  Privacy and confidentiality will be protected using de-identification of all individual-level data. Audio recordings and transcripts will not be shared so as to maintain participant privacy.
Time Frame: The scientific dataset will be shared at the time of associated publications and will be made available for as long as it is useful to the larger research community (i.e., in perpetuity).
Access Criteria: All individual-level data sets will be shared in openICPSR.

REFERENCES:
- [Derived] Giordano NA, Kaplan DM, Peacock C, Vyas I, Pozzo N, Shelton M, Escoffery C, Rana S, Raison CL, Grant GH, Mascaro JS. Protocol to examine the feasibility and acceptability of a randomized controlled trial of a chaplain-delivered compassion intervention to improve psychological safety among interprofessional healthcare teams. Pilot Feasibility Stud. 2025 Nov 13;11(1):141. doi: 10.1186/s40814-025-01712-7. PMID 41258216